CLINICAL TRIAL: NCT07348926
Title: Examination of Families' Psychological Status and Quality of Life According to the Functional Independence Status of Children With Rare Genetic Diseases in Early Childhood
Brief Title: The Relationship Between Functional Independence and Family Well-being in Children With Rare Genetic Disorders
Status: Recruiting | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Yağmur Erkan, Graduate Student Researcher, Bahçeşehir University
Other Study IDs: BAU-FTR-YE-01
Record Dates: First submitted 2025-12-11; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Rare Genetic Disorders; Quality of Life; Functional Impairment
Keywords: Rare Genetic Disorders; physical therapy; Depression; Quality of Life; Family
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lower Functional Independence: Children with rare genetic disorders whose functional independence level is lower based on the Pediatric Functional Independence Measure (WeeFIM). Caregivers of these children are included in the study.
- Higher Functional Independence: Children with rare genetic disorders whose functional independence level is higher based on the Pediatric Functional Independence Measure (WeeFIM). Caregivers of these children are included in the study.

SUMMARY:
This study aims to examine the psychological status and quality of life of families with children who have rare genetic disorders. The focus of the study is to understand how the child's level of functional independence relates to the well-being of the family. Functional independence will be assessed using standardized tools, and parental psychological status and quality of life will be evaluated with validated questionnaires.

The information gathered from this study may help improve the understanding of how rare genetic disorders affect family dynamics and daily functioning. The results may guide health care professionals in planning family-centered physiotherapy, psychological support, and care programs.

DETAILED DESCRIPTION:
This observational, descriptive, and cross-sectional study aims to examine the associations between the functional independence levels of young children diagnosed with rare genetic disorders and various psychosocial outcomes of their caregivers, including depression, family functioning, sleep quality, and overall quality of life. Rare genetic disorders often begin in early childhood, require long-term medical follow-up and rehabilitation, and may negatively affect both the daily routines and psychosocial well-being of families. In this context, understanding family-centered physiotherapy and its role as a protective factor is crucial for strengthening family systems and supporting rehabilitation success.

The study population consists of caregivers of children aged 0-4 years with rare genetic diagnoses who are receiving physiotherapy at a rehabilitation center in Istanbul. A sample size of 45 participants was calculated based on Cohen's effect size approach, assuming a medium effect size (d = 0.5).

Functional independence of the child will be assessed using the Pediatric Functional Independence Measure (WeeFIM). Based on WeeFIM scores, parents will be categorized into two groups according to the child's functional level. Caregiver depression levels will be assessed using the Beck Depression Inventory; family functioning will be evaluated with the Family Functionality in Rehabilitation Scale; family impact will be measured with the Family Impact Scale; sleep quality will be evaluated using the Pittsburgh Sleep Quality Index; and quality of life will be assessed using the Nottingham Health Profile. Demographic information and details of physiotherapy participation will also be collected.

Data collection will begin after ethical approval and will last approximately three months. Following informed consent, all participants will complete the questionnaires in Turkish. The findings of this study are expected to provide a comprehensive understanding of the multidimensional challenges faced by families of children with rare genetic disorders and may guide the development of family-centered physiotherapy, psychosocial interventions, and supportive care programs.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children aged 0-4 years diagnosed with a rare genetic disorder.
* The child must have been receiving physiotherapy for at least 6 months.
* Caregivers who voluntarily agree to participate and provide informed consent.
* Caregivers who are able to read and understand Turkish to complete the questionnaires.

Exclusion Criteria:

* Caregivers who have cognitive or language limitations that prevent them from completing the questionnaires.
* Caregivers who decline participation or submit incomplete questionnaire forms.
* Children or caregivers with an additional medical or neurological condition that prevents participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of caregivers of children aged 0-4 years who have been diagnosed with rare genetic disorders and receive physiotherapy services at a rehabilitation center in Istanbul, Turkey. Participants are primary caregivers responsible for the child's daily care and able to complete Turkish-language questionnaires. The population reflects a clinical sample receiving ongoing rehabilitation, rather than a community-based or general population sample
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Level of the Child (WeeFIM) | At baseline (study enrollment)
  The functional independence level of children with rare genetic disorders will be assessed using the Pediatric Functional Independence Measure (WeeFIM). This scale evaluates functional abilities in self-care, mobility, and cognition. Higher scores indicate greater functional independence.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | At baseline (study enrollment)
  Caregiver depressive symptoms will be assessed using the Beck Depression Inventory (BDI). This scale measures emotional, cognitive, and physical symptoms of depression. Higher scores indicate higher levels of depressive symptoms.eck Depression Inventory (BDI), higher scores indicate greater severity of depressive symptoms.
Family Functionality in Rehabilitation | At baseline (study enrollment)
  This outcome will assess the caregiver's perceived role and functionality in the child's rehabilitation process using the Family Functionality in Rehabilitation Scale. Higher scores indicate better family functioning within the rehabilitation setting.
Family Impact (Family Impact Scale) | At baseline (study enrollment)
  The Family Impact Scale will be used to evaluate how the child's rare genetic condition affects family routines, emotional well-being, and daily functioning. Higher scores indicate greater perceived impact on family life.
Sleep Quality (Pittsburgh Sleep Quality Index - PSQI) | At baseline (study enrollment)
  Caregiver sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI), which evaluates sleep duration, latency, disturbances, and overall sleep quality. Higher scores reflect poorer sleep quality.
Quality of Life (Nottingham Health Profile - NHP) | At baseline (study enrollment)
  Caregiver quality of life will be assessed using the Nottingham Health Profile (NHP), which evaluates emotional, social, and physical domains of well-being. Higher scores indicate poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğçe Tahmaz, PhD, Principal Investigator — Bahçeşehir University
Locations (1):
- Bahcesehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No